CLINICAL TRIAL: NCT04168060
Title: The Effect of Routine Crura Dissection in Sleeve Gastrectomy on Post-Operative Symptoms
Brief Title: Crural Dissection in Sleeve Gastrectomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Changes in practice patterns. From COVID-related disruptions to the adoption of ERAS protocols and robotic surgery, there was significant variability in standards of care making direct comparison between groups impractical.
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Nestor De La Cruz-Munoz, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20190190
Record Dates: First submitted 2019-11-15; First posted 2019-11-19 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Sleeve Gastrectomy
Keywords: sleeve gastrectomy; crura dissection; bariatric surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Crura Dissection (Experimental): Participants with a visually detectable hiatal hernia at the time of sleeve gastrectomy procedure will undergo a crura dissection and hiatal hernia repair.
  Interventions: Procedure: Crura dissection; Procedure: Sleeve gastrectomy; Procedure: Hiatal hernia repair
- National Practice (Experimental): Participants with no detectable hiatal hernia will be randomized to either Group 2 or 3. Group 2 participants will be treated to the national practice patterns of complete dissection of the curvature of the stomach without dissection of the crura.
  Interventions: Procedure: Sleeve gastrectomy
- Standard of Care (Experimental): Participants with no detectable hiatal hernia will be randomized to either Group 2 or 3. Group 3 participants will undergo the institutional standard of care with the dissection of the crura.
  Interventions: Procedure: Crura dissection; Procedure: Sleeve gastrectomy

INTERVENTIONS:
Procedure: Crura dissection — The diaphragmatic crura, one of two tendon structures below the diaphragm, will be removed during the laparoscopic sleeve gastrectomy.
  Arms: Crura Dissection; Standard of Care
Procedure: Sleeve gastrectomy — Surgical weight-loss procedure in which the stomach is reduced to about 15% of its original size, by surgical removal of a large portion of the stomach along the greater curvature.
Procedure: Hiatal hernia repair — This involves tightening the opening in your diaphragm with stitches to keep your stomach from bulging upward through the opening in the muscle wall.
  Arms: Crura Dissection

SUMMARY:
The purpose of this study is to identify if there is a benefit in routine dissection of the diaphragmatic crura during sleeve gastrectomy.

ELIGIBILITY:
Inclusion criteria:

1. All patients undergoing primary sleeve gastrectomy at the University of Miami Division of Bariatric surgery
2. Age between 18-69 years
3. Able to provide consent

Exclusion criteria:

1. History of anti-reflux procedure
2. History of foregut surgery
3. Narcotic dependence
4. History of gastroparesis
5. Special/vulnerable populations such as minors, patients unable to consent, pregnant women, and prisoners will not be included in the study

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
Change in Perioperative Symptoms as assessed by the Intermediate and Late-Post Operative Pain, Nausea and Dysphagia Questionnaire | Day 1, 12 months
  The Intermediate and Late Post-Operative Pain, Nausea and Dysphagia Questionnaire is a 7-item questionnaire with scores ranging 0-40 with the higher score indicating severe symptoms.
Change in Perioperative Symptoms as assessed by the Rhodes Index of Nausea, Vomiting and Retching Questionnaire | Day 1, 12 months
  The Rhodes Index of Nausea, Vomiting and Retching Questionnaire is an 8-item questionnaire with scores ranging from 0 to 32 with a higher score indicating increased symptoms of nausea.
Change in Perioperative Symptoms as assessed by the Gastroesophageal Reflux Disease-Questionnaire (GERD-Q) | Baseline, 12 months
  The GERD-Q has a scoring range between 0-18 with a higher score indicating increased likelihood of GERD.
Change in Perioperative Symptoms as assessed by the Brief Esophageal Dysphagia Questionnaire (BEDQ) | Baseline, 12 months
  The BEDQ has a scoring range between 0-40 with a higher score indicating increased symptoms of dysphagia.

SECONDARY OUTCOMES:
Correlation of the presence of hiatal hernias | Day 1
  Correlation of the presence of hiatal hernias between pre-operative upper Gastrointestinal (GI) series and surgical findings.

CONTACTS AND LOCATIONS:
Overall Officials: Nestor De La Cruz-Munoz, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Medical Campus, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No